CLINICAL TRIAL: NCT04447300
Title: Outcomes of High Power Application in Catheter Ablation of Paroxysmal Atrial Fibrillation Guided by Unipolar Signal Modification.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Abdelrady Abdelsalam Farghaly, Assistant lecturer of cardiovascular medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: atrial fibrillation ablation
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Atrial fibrillation ablation - unipolar signal modification
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard power application (Active Comparator)
  Interventions: Procedure: Standard power application
- High power application (Active Comparator)
  Interventions: Procedure: high power application

INTERVENTIONS:
Procedure: high power application — Radiofrequency delivery was performed in a point-by point fashion and continuously (an inter-lesion distance of 6 mm) with 50 W and 70 W and the ablation time for each point is limited to 7s and repeated if needed till the Unipolar signal modification turn to complete positive R wave.
  Arms: High power application
Procedure: Standard power application — Standard power application
  Arms: Standard power application

SUMMARY:
Pulmonary vein isolation (PVI) is the cornerstone of catheter ablation procedures in patients with paroxysmal atrial fibrillation (PAF) [1]. However, the incidence of atrial fibrillation (AF) recurrence remains high [2], mostly due to pulmonary vein (PV) reconnection [1], emphasizing the formation of transmural lesions to achieve complete conduction block along the ablation lines [3].

Previous studies have shown that elimination of the negative component of the unipolar electrogram (UP-EGM) during radiofrequency applications reflects transmural lesions. The persistence of such a negative component consistently corresponds to non-trans mural lesions [4].

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) is the cornerstone of catheter ablation procedures in patients with paroxysmal atrial fibrillation (PAF) [1]. However, the incidence of atrial fibrillation (AF) recurrence remains high [2], mostly due to pulmonary vein (PV) reconnection [1], emphasizing the formation of transmural lesions to achieve complete conduction block along the ablation lines [3].

Previous studies have shown that elimination of the negative component of the unipolar electrogram (UP-EGM) during radiofrequency applications reflects transmural lesions. The persistence of such a negative component consistently corresponds to non-trans mural lesions [4].

The high-power short duration (HPSD) RF application applies to all RF energies delivered at more than 40 W [5]. Higher the power more is the resistive heating causing wider tissue injury [5]. The lesion size with HPSD is larger in width but lesser in depth compared to lower powers with longer duration [5]. In contrast, RF applications of lower power and longer duration result in larger dissipation of RF energies deep into the tissues due to conductive heating causing tissue destruction at greater depths [6]. Hence, there is a risk of collateral tissue damage [5].

HPSD ablation has been advocated as a means to minimize the risk of collateral organ damage as the lesions are smaller in depth. However, Maintaining a high power for a constant duration in the absence of a guide may not be the right strategy [5].

Unipolar waveform modification by complete elimination of the negative component may serve as a guide for HPSD ablation [5].

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation

Exclusion Criteria:

* Age< 18 or > 80 years old,
* Atrium (LA) diameter > 50 mm,
* The presence of a mechanical mitral valve prosthesis,
* Left ventricular ejection fraction < 40%,
* Abnormal thyroid function,
* Contraindication to anticoagulant therapy,
* Current malignancy,
* Prior catheter or surgical AF ablation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Ablation success at 6-month after the index procedure | 6 months
  Ablation success is defined as no recurrence with no anti-arrhythmic drugs by taking history of symptoms from the patient and by Holter 48 Hours.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kottmaier M, Popa M, Bourier F, Reents T, Cifuentes J, Semmler V, Telishevska M, Otgonbayar U, Koch-Buttner K, Lennerz C, Bartkowiak M, Kornmayer M, Rousseva E, Brkic A, Grebmer C, Kolb C, Hessling G, Deisenhofer I. Safety and outcome of very high-power short-duration ablation using 70 W for pulmonary vein isolation in patients with paroxysmal atrial fibrillation. Europace. 2020 Mar 1;22(3):388-393. doi: 10.1093/europace/euz342. PMID 31872249